CLINICAL TRIAL: NCT06087965
Title: Efficacy and Safety of Fingolimod in Minimal Invasive Treatment of Intracerebral Hemorrhage
Brief Title: Fingolimod in Minimal Invasive Treatment of Intracerebral Hemorrhage
Acronym: FMIICH
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202307-11
Record Dates: First submitted 2023-10-09; First posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Intracerebral Hemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage | interventions — Fingolimod Hydrochloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fingolimod group (Experimental): 0.5mg/day oral fingolimod over a course of 3 consecutive days
  Interventions: Drug: Fingolimod
- Control group (No Intervention): No fingolimod will be administered.

INTERVENTIONS:
Drug: Fingolimod — 0.5mg/day oral fingolimod over a course of 3 consecutive days
  Arms: Fingolimod group

SUMMARY:
Intracerebral hemorrhage (ICH) is a critical disease of public health importance. Inflammatory mechanisms play a significant role in ICH. Thus, immune targets are supposed to be effective in protecting the neurological function of ICH. Fingolimod, a sphingosine-1-phosphate receptor regulator (FTY720), is an effective immunology modulator. It has been widely used in autoimmune disease and has also been testified effective in ICH who received conservative treatment. The present study aims to evaluate the efficiency and safety of fingolimod for ICH with minimal invasive treatment.

DETAILED DESCRIPTION:
40 ICH patients who meet the inclusion criteria will be enrolled in the present study.

All ICH patients will be screened. If meeting the including criteria, the investigators will contact the family, explain the study, and send a consent form for review.

After obtaining written consent from the family, patients randomly assigned to the fingolimod group will be given 0.5mg/day oral fingolimod over a course of 3 consecutive days. Patients assigned to the control group will not receive fingolimod. All patients will receive minimal invasive puncture and drainage of hematoma. The investigators will evaluate the neurofunctional before and 30 days, 90 days and 180 days after oral fingolimod. CT scan will be performed at before, 7 and 14 days after oral fingolimod. 5ml intravenous blood for flow cytometry is also taken before and 1day, 3days, 7days after fingolimod use.

ELIGIBILITY:
Inclusion Criteria:

* spontaneous basal ganglia ICH with volume larger than 20ml;
* age: 18-80 years;
* admission Glasgow Coma Scale score: 5-12;
* admitting to hospital with 24 hours after injury;
* no fever or signs infection on admission to hospital;
* admission heart rate≥60/min on admission.

Exclusion Criteria:

* refuse follow-up;
* received operation before admitting to hospital;
* hemorrhage by tumor, arteriovenous malformation, arterial aneurysm, hematological disease or traumatic brain injury;
* severe vomiting;
* mRS>1 before ICH;
* prior history of bradycardia;
* prior history of Atrioventricular block;
* prior history of traumatic brain injury, craniotomy or stroke;
* expected lifetime less than 1 year;
* undergoing antitumor, antiepileptic, immunomodulatory or immunosuppressive therapy;
* admitting to other ongoing study;
* systemic disease: uremia, liver cirrhosis, malignant tumor, mental disease, drug or alcohol dependence;
* received anticoagulant or antiplatelet therapy within 7 days;
* intraventricular hemorrhage requires intraventricular catheterization.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-10-11 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
modified Rankin Scale | 90 days and 180 days after ICH
  Neurological outcome, range: 0-6. The higher scores mean a worse outcome.

SECONDARY OUTCOMES:
The National Institutes of Health Stroke Scale | 90 days and 180 days after ICH
  Neurological outcome, range: 0-42. The higher scores mean a worse outcome.
Modified Barthel Index | 90 days and 180 days after ICH
  Neurological outcome, range: 0-100. The higher scores mean a better outcome.
Montreal Cognitive Assessment Scale | 90 days and 180 days after ICH
  Neurological outcome, range: 0-30. The higher scores mean a better outcome.
Volume of perihematomal edema | Baseline on admission, 7 days and 14 days after ICH
  Volume of perihematomal edema measured on head Computerised Tomography

CONTACTS AND LOCATIONS:
Overall Officials: Yan Qu, Study Chair — Tang-Du Hospital

IPD SHARING:
Plan to Share IPD: Yes
the baseline characteristic, treatments and functional outcomes will be shared with other researchers
Supporting Information: Study Protocol, CSR
Time Frame: the data will be available after the study is finished for 3 years
Access Criteria: Individual participant data will be shared on a website available to other researchers.